CLINICAL TRIAL: NCT03842709
Title: Non-opioid Pramipexole Suppresses Immune NLRP3 Reactivity for Pain Control
Brief Title: Non-Opioid Pramipexole and Pain
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Erin Damita Milligan, Associate Professor, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18-592
Record Dates: First submitted 2019-02-08; First posted 2019-02-15 (Actual); Results first posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Pramipexole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Treatment + Placebo (Placebo Comparator): Patients reporting sub-optimal results of pain therapy, assigned to placebo in addition to routine care.
  Interventions: Other: Placebo
- Standard Treatment + Pramipexole (Experimental): Patients reporting sub-optimal results of pain therapy, assigned to receive pramipexole in addition to routine care.
  Interventions: Drug: Pramipexole Oral Tablet

INTERVENTIONS:
Drug: Pramipexole Oral Tablet — Initial dosage of 0.125 mg pramipexole daily, potentially titrated upward in 0.125 increments to a maximum of 0.5 mg daily, for 4 weeks.
  Arms: Standard Treatment + Pramipexole
Other: Placebo — Administration of placebo
  Arms: Standard Treatment + Placebo

SUMMARY:
The long-term goal of this proposal is to identify non-opioid drugs that harness endogenous anti-inflammatory mechanisms resulting in the suppression of proinflammatory cytokines such as IL-1ß providing a novel approach to treat chronic pain in people while lacking potential for addictive side effects.

Specific Aim I: pramipexole blocks the activation of NLRP3 and consequent production and release of the proinflammatory cytokines IL-1ß, IL-6 and TNF-α, and increases production of the anti-inflammatory cytokine interleukin-10 (IL-10).

The goal of Aim I (Phase I) experiments is to examine the specific anti-inflammatory mechanisms of pramipexole on PAMP, DAMP and opioid stimulated immune cells, THP-1 cells will be used.

Specific Aim II: pramipexole treatment will provide therapeutic benefit to patients experiencing suboptimal pain relief from current standard therapy with concurrent reduction of TLR4-NLRP3-cytokine expression in peripheral blood mononuclear cells.

The goal of Aim II (Phase II) will be to determine the therapeutic benefit of pramipexole for pain, which is a repurposing of this FDA-approved drug with a good safety profile.

1.2. Our overarching hypothesis is that pramipexole will control clinical pain by suppressing the activation of the TLR4-NLRP3-IL-1ß pathway and prevent IL-1ß release from peripheral immune cells. These findings have provided the current impetus to examine pain therapeutic drugs targeting immune-related factors either upstream or downstream of IL-1ß signaling.

DETAILED DESCRIPTION:
The long-term goal of this proposal is to identify non-opioid drugs that harness endogenous anti-inflammatory mechanisms resulting in the suppression of proinflammatory cytokines such as IL-1ß providing a novel approach to treat chronic pain in people while lacking potential for addictive side effects.

This study is conducted to determine the therapeutic benefit of pramipexole for pain, which is a repurposing of this FDA-approved drug with a good safety profile. In collaboration with Dr. Koshkin (co-I at UNMH Pain Clinic), patients from the UNM pain clinic will be recruited who are experiencing modest or suboptimal pain relief. The patient will meet the CTSC Clinical Research Coordinator, who will escort the patient to the Clinical Research Lab. At the time, an explanation of the study, consent, the Brief Pain Inventory survey will be completed, blood draw and Clincard will be given to the patient ($15/visit). Scheduling for the midterm visit to the CTSC (at the end of two weeks) will be determined. At the time of consent, all patients will be under standard pain treatment and will be randomized into two groups: (1) patients receiving pramipexole in addition to their standard ongoing pain treatment, or (2) no pramipexole but will continue to receive the standard pain treatment. Patients will be followed up in the morning at weekly intervals to provide pain scores either by phone (for week 1 and 3), or by return visit (for end of week 2 and at the end of week 4) until study termination which is at the end of week 4.. At the initiation of the study and at the end of 4 weeks, blood will be collected and analyzed for mRNA for TLR4, p38, NFkB, NLRP3-ASC, Caspase-1, IL-1ß, TNF-α, HMGB1, and IL-10. The dose and route of administration of pramipexole will be identical to that previously approved for the treatment of Restless Legs Syndrome and according to manufacturer's recommended prescribing protocol (Mirapex, Boehringer Ingelheim Int. GmbH). Briefly, oral dosage will be titrated each week to achieve a weekly total daily dose of 0.125 (mg), 0.250, or 0.5. Patients will take one capsule containing pramipexole of placebo 2-3 hours before bedtime.

Patient recruitment, assessment of Brief Pain Inventory (BPI): Pain scores and blood draws will be conducted at the CTSC Participant Clinical Interactions Unit with the CTSC Clinical Research Coordinator. Blood samples collected by the CTSC Clinical Research Coordinator will be analyzed at the Center for Molecular Discovery by personnel from Dr. Milligan's lab, trained by personnel from the Center for Molecular Drug Discovery (Director; Dr. Sklar, co-I). Personnel from the Milligan lab have expertise in inflammatory marker analysis from PBMCs [57, 58]. All freshly collected blood samples will be frozen and stored by the Clinical Research Coordinator at the CTSC Clinical Laboratory and will be transported to the Center for Molecular Drug Discovery once ALL of the samples for the study have been collected for mRNA and protein analysis. This is to allow for assay to be conducted at the same time to avoid potential effect of 'time of assay' that may impact data.

All subjects will therefore meet with the CTSC Clinical Research Coordinator for a total of 3 times; at the initiation of the study, at mid-term when the second batch of drug is dispensed and unused drug is returned, and at termination for a second and final blood draw and providing all completed Brief Pain Inventory surveys (4/patient). At the termination of the study, patients will turn in their paper copies of the Brief Pain Inventory questionnaire completed for each week of the study (total 4 weeks). Original data records are important to demonstrate all necessary physical documentation of the study.

The long-term goal of this proposal is to identify non-opioid drugs that harness endogenous anti-inflammatory mechanisms resulting in the suppression of proinflammatory cytokines such as IL-1ß providing a novel approach to treat chronic pain in people while lacking potential for addictive side effects.

ELIGIBILITY:
Inclusion Criteria:

* Nonmalignant chronic pain patients at University of New Mexico Pain Clinic, reporting suboptimal pain control, who state an interest to try something new to improve pain relief
* Pain score of 5 or greater (0-10 scale)
* Pain lasting more than 3 months

Exclusion Criteria:

* Patients who do not speak English or Spanish
* Patients unable to consent
* Women who are not post-menopausal, or who have not undergone an oophorectomy/hysterectomy
* Patients who have chronic pulmonary, kidney or liver disease
* Patients with a body mass index (BMI) ≥35
* Patients with a cancer diagnosis within the last 2 years (except non-melanoma skin cancer)
* Patients who are currently lactating
* Patients with a history of orthostatic hypotension
* Patients diagnosed with a dissociative disorder
* Patients with Parkinson's disease, and/or currently taking dopamine agonist prescription medications
* Prisoners and other institutionalized individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2021-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin D Milligan, PhD, Principal Investigator — University of New Mexico Health Sciences Center (HSC)
Locations (1):
- University of New Mexico Hospital, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Treatment + Placebo | Standard Treatment + Pramipexole
Started | 7 | 6
Initiated Treatment | 6 | 5
Completed | 3 | 3
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: 2 participants at enrollment did not complete the Pain Inventory questionnaire, and were withdrawn from the study very early in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Treatment + Placebo | Standard Treatment + Pramipexole | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 3 | 2 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11
Pain scores at enrollment [Mean (Standard Deviation); unit: units on a scale] — Brief Pain Inventory scale rating the worst pain within previous 24 hrs; 0 = no pain, and 10 = worst pain.
  units on a scale | 7.5 (2.0) | 8.2 (1.8) | 7.8 (1.8)
Blood cytokine levels at enrollment (IL-1b) [Mean (Standard Deviation); unit: Fold change from baseline] — Measures a "fold increase" in expression relative to housekeeping-gene baseline.
  Fold change from baseline | 7.5 (3.1) | 13.9 (7.5) | 10.7 (6.4)

OUTCOME MEASURES:

1. Primary Outcome: Brief Pain Inventory Score
Description: Change in self-reported effect of pain on quality of life. The "Brief Pain Inventory, Short Form," instrument will be used. It records severity (0-10 scale; 10= worst pain) at its worst.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Treatment + Placebo | Standard Treatment + Pramipexole
Number analyzed (Participants) | 3 | 3
score on a scale | 8 (1) | 6.7 (3.2)

2. Secondary Outcome: mRNA Results IL-1b
Description: Fold change of the mRNA gene expression from the house keeping gene and the controls.
Time Frame: 4 weeks
Population: Four participants did not provide relevant blood samples.
Measure: Mean (Standard Deviation); unit: Fold change
Arm/Group | Standard Treatment + Placebo | Standard Treatment + Pramipexole
Number analyzed (Participants) | 4 | 3
Fold change | 16.1 (8.1) | 8.6 (8.6)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Standard Treatment + Placebo | Standard Treatment + Pramipexole
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Treatment + Placebo (N=6) | Standard Treatment + Pramipexole (N=5)
dizziness (Nervous system disorders) | 0 (0) | 1 (1) — experienced a single fall

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/09/NCT03842709/Prot_SAP_001.pdf
  • Informed Consent Form (2018-11-09): https://cdn.clinicaltrials.gov/large-docs/09/NCT03842709/ICF_000.pdf